CLINICAL TRIAL: NCT07025837
Title: The Effects of an LED Face Mask & Neck and Chest Mask On Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freedom Laser, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20679
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Skin Aging; Sun Damaged Skin
Keywords: Skin Health; Neck and Chest Mask

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iRESTORE Illumina LED Device Group (Experimental): All participants will use the iRESTORE LED Face Mask and Neck & Chest Mask daily for 10 minutes each night. For the face mask, Mode 1 will be used.
  Interventions: Device: iRESTORE Illumina LED Face Mask and Neck & Chest Mask

INTERVENTIONS:
Device: iRESTORE Illumina LED Face Mask and Neck & Chest Mask — A pair of light-emitting diode (LED) therapy devices designed for at-home use. The facial and neck/chest masks deliver low-level red light therapy through embedded LEDs to improve visible signs of skin aging.

SUMMARY:
This 12-week single-group virtual study evaluates the effects of the iRESTORE Illumina LED Face Mask and Neck & Chest Mask on skin health in adult females. Participants will use the devices daily for 10 minutes and complete scheduled surveys and photographs to assess improvements in skin appearance via both dermatologist assessment and participant perception.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 25-55 years.
* Willing to follow the study protocols.
* Self-reported issues with at least two of the following: Fine lines, Wrinkles, Hyperpigmentation, Dark spots, Reduced elasticity
* Self-report concerns with at least one of the following: Crepey skin on the neck and chest, Sun damage on neck and chest
* Willing to avoid introducing any new products, prescription medications, or supplements that target skin health during the study period.
* If taking oral supplements or herbal remedies targeted at skin health and appearance, have been consistently taking these for at least 3 months prior to starting the study.
* Is willing to maintain the routine of any oral supplements or herbal remedies targeted at skin health and appearance for the duration of the study.
* Has been using the same skincare routine for at least one month prior to the study start date.
* Willing to maintain the same skincare routine and products throughout the study.
* Willing to avoid direct sun exposure during the study duration
* Willing to wear sunscreen if have to be in the sun

Exclusion Criteria:

* Anyone who is extremely satisfied with their skin.
* Anyone who has any chronic health conditions such as oncological (cancer) or psychiatric disorders.
* Anyone who is planning to undergo facial treatments during the study period, including botox, dermal filler, chemical peels, etc. or has experienced any of these treatments in the last 3 months.
* Anyone diagnosed with a skin condition affecting the face and/or neck who has had an active flare-up or breakout within the last year. This includes but is not limited to acne, eczema, psoriasis, rosacea, seborrheic dermatitis, vitiligo, urticaria (hives), warts, atopic dermatitis, melasma, and contact dermatitis.
* Currently using any prescription medications that may affect the skin condition including but not limited to the following:
* Corticosteroids like prednisone, methylprednisolone
* Antipsychotics like olanzapine (Zyprexa), risperidone (Risperdal), quetiapine (Seroquel)
* SSRIs and SNRIs like fluoxetine (Prozac), sertraline (Zoloft), venlafaxine (Effexor)
* Anticonvulsants like phenytoin (Dilantin), lamotrigine (Lamictal), and carbamazepine (Tegretol)
* Antihypertensives like lisinopril (Zestril), amlodipine (Norvasc), and propranolol (Inderal)
* Antithyroid medications like Tapazole (methimazole), Propyl-Thyracil (propylthiouracil)
* Anyone with a history of skin cancer or precancerous skin lesions on the face.
* Anyone who has any known serious allergic reactions that require the use of an Epi-Pen.
* Anyone who has any known allergies to ingredients commonly found in skincare products.
* Anyone who is pregnant, breastfeeding, or trying to conceive
* Anyone who cannot/will not commit to the study protocol.
* Anyone with a history of substance abuse.
* Anyone who has undergone an invasive medical procedure in the three weeks prior to the study or has a procedure planned during the study duration.
* Anyone with a known allergic reaction to aluminum or plastics.
* Anyone who suffers from any photosensitive disorder (sensitization to light).
* Anyone with uncontrolled acne.
* Anyone taking any prescription medication, over-the-counter supplements, or herbal supplements regularly (three or more days per week) that can cause photosensitivity including but not limited to the following:
* Antibiotics like tetracyclines (e.g., doxycycline, tetracycline) or sulfonamides (e.g., Bactrim), fluoroquinolones (e.g., ciprofloxacin, levofloxacin)
* Antifungals like Griseofulvin or Vfend (voriconazole)
* Diuretics like drugs ending in -thiazides
* NSAIDs like ibuprofen and Aleve (naproxen)
* Retinoids or Vitamin A (e.g., Accutane (isotretinoin), (Retin-A) tretinoin
* Antidepressants (e.g., SSRIs, Elavil (amitriptyline), Tofranil (imipramine)
* Antihistamines like Phenergan (promethazine)
* Antimalarial medications
* Statins like Lipitor (atorvastatin), Zocor (simvastatin)
* Antiarrhythmics like Pacerone (amiodarone)
* St. John's wort
* Anyone who suffers from light-induced headaches or migraines.
* Anyone with a medical history of seizures or epilepsy triggered by light.
* Anyone with an electronic implanted device such as a defibrillator, neurostimulator, pacemaker, or ECG monitor.
* Anyone with a known history of carotid artery disease, stroke or transient ischemic attack (TIA), carotid stenosis, unstable blood pressure, easy fainting, thyroid disease, or of individuals about to undergo surgical procedures in the neck area.
* Anyone who has stopped hormonal birth control in the past month.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | iRESTORE Illumina LED Device Group
Started | 38
Completed | 36
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Age, Customized [Count of Participants; unit: Participants]
  25 to 55 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reported as Having an Improvement in Overall Skin Health as Evaluated by Dermatologist Grading
Description: Participants will submit photos, which are reviewed by dermatologists using a standardized grading system to evaluate visible changes in overall skin health.
Time Frame: Baseline, Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 36
Participants | 29

2. Primary Outcome: Percentage of Participants Reported as Having an Improvement in Fine Lines and Wrinkles as Evaluated by Dermatologist Grading
Description: Participants will submit photos, which are reviewed by dermatologists using a standardized grading system to evaluate visible changes in fine lines and wrinkles.
Time Frame: Baseline, Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 36
Participants | 17

3. Primary Outcome: Percentage of Participants Reported as Having an Improvement in Skin Pigmentation as Evaluated by Dermatologist Grading
Description: Participants will submit photos, which are reviewed by dermatologists using a standardized grading system to evaluate visible changes in skin pigmentation.
Time Frame: Baseline, Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 36
Participants | 24

4. Primary Outcome: Percentage of Participants Reported as Having an Improvement in Skin Redness as Evaluated by Dermatologist Grading
Description: Participants will submit photos, which are reviewed by dermatologists using a standardized grading system to evaluate visible changes in skin redness.
Time Frame: Baseline, Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 36
Participants | 26

5. Primary Outcome: Percentage of Participants Reported as Having an Improvement in Signs of Aging as Evaluated by Dermatologist Grading.
Description: Participants will submit photos, which are reviewed by dermatologists using a standardized grading system to evaluate visible changes in signs of aging.
Time Frame: Baseline, Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 36
Participants | 24

6. Secondary Outcome: Self-Reported Improvement in Overall Skin Hydration
Description: This outcome measures the change in participant-reported scores for overall skin hydration from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale for skin hydration, including Extremely Dry (=1), Mildly Dry (=2), Neither dry nor hydrated (=3), Hydrated with room for improvement (=4), and Optimally hydrated (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: The number of participants analyzed at each time point reflects the available data from participants who completed assessments at that specific time point. The decreasing numbers are due to participant dropouts and missed measurements. All data were analyzed using an intention-to-treat (ITT) approach, with results reported for all participants who provided data at each respective time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.74 (0.98)
  Week 2 | 3.05 (1.18)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.97 (1.09)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.14 (1.00)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.46 (1.12)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.35 (1.11)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 3.59 (1.09)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p > 0.9999, ANOVA — Week 2 compared to the baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p > 0.9999, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.6342, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0231, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0862, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0033, ANOVA — Week 12 compared to baseline

7. Secondary Outcome: Self-Reported Improvement in Skin Plumpness
Description: This outcome measures the change in participant-reported scores for skin plumpness from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of plumpness, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.97 (0.75)
  Week 2 | 3.21 (0.84)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.51 (0.73)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.76 (0.64)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.76 (0.64)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.86 (0.63)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4.05 (0.62)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.1176, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0030, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0001, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline

8. Secondary Outcome: Self-Reported Improvement in Skin Tone
Description: This outcome measures the change in participant-reported scores for skin tone from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale for skin tone, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.79 (0.78)
  Week 2 | 3.05 (0.96)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.43 (0.77)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.62 (0.76)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.92 (0.68)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.89 (0.66)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4.08 (0.68)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.9751, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0078, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0003, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

9. Secondary Outcome: Self-Reported Improvement in Skin Texture
Description: This outcome measures the change in participant-reported scores for skin texture from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of skin texture, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.92 (0.94)
  Week 2 | 3.32 (0.84)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.57 (0.69)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.73 (0.69)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.86 (0.75)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.95 (0.57)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4.19 (0.57)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0544, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0036, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0001, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to Baseline

10. Secondary Outcome: Self-Reported Improvement in Facial Skin Glow
Description: This outcome measures the change in participant-reported scores for facial skin glow from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of facial skin glow, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.50 (0.89)
  Week 2 | 3.26 (1.00)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.57 (0.77)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.81 (0.66)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.81 (0.74)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.92 (0.64)
  Week 12 | 4.16 (0.65)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0001, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

11. Secondary Outcome: Self-Reported Improvement in Facial Skin Health
Description: This outcome measures the change in participant-reported scores for facial skin health from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of facial skin health, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 3.05 (0.90)
  Week 2 | 3.42 (1.00)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.68 (0.63)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.81 (0.62)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.76 (0.68)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.89 (0.61)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4.16 (0.65)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.1438, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0092, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0003, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0015, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

12. Secondary Outcome: Self-Reported Improvement in Facial Skin Appearance
Description: This outcome measures the change in participant-reported scores for facial skin appearance from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of facial skin appearance, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.79 (0.84)
  Week 2 | 3.26 (1.03)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.51 (0.69)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.70 (0.70)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.86 (0.75)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.92 (0.68)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4.08 (0.68)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0041, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0001, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

13. Secondary Outcome: Self-Reported Improvement in Skin Tone Evenness.
Description: This outcome measures the change in participant-reported scores for skin tone evenness from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of skin tone evenness, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.50 (0.83)
  Week 2 | 2.97 (0.97)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.35 (0.75)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.46 (0.80)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.70 (0.81)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.97 (0.76)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4.00 (0.82)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0249, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

14. Secondary Outcome: Self-Reported Improvement in Facial Skin Clarity
Description: This outcome measures the change in participant-reported scores for facial skin clarity from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of facial skin clarity, including Very bad (=1), Bad (=2), Neither good nor bad (=3), Good (=4), and Very good (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 3.16 (1.13)
  Week 2 | 3.26 (1.13)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.59 (0.86)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.70 (0.94)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.92 (0.89)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.92 (0.92)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4.14 (0.86)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p > 0.9999, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.7453, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.2118, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0111, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0150, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0003, ANOVA — Week 12 compared to baseline

15. Secondary Outcome: Self-Reported Improvement in Lift and Firmness of Skin
Description: This outcome measures the change in participant-reported scores for lift and firmness of skin from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of skin lift and firmness, including Not at all (=1), A little bit (=2), Somewhat (=3), Very much (=4), and Extremely (=5). Higher scores indicate greater improvement. This is a positively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.29 (0.73)
  Week 2 | 2.76 (0.88)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 3.05 (0.70)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 3.11 (0.70)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 3.46 (0.80)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 3.46 (0.90)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 3.57 (0.90)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0199, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

16. Secondary Outcome: Self-Reported Improvement in the Severity of Skin Redness
Description: This outcome measures the change in participant-reported scores for severity of skin redness from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of skin redness severity, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.55 (0.89)
  Week 2 | 2.37 (0.71)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.22 (0.67)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 2.27 (0.61)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 2.03 (0.69)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 2.00 (0.71)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 1.89 (0.77)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.4438, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0412, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0943, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0017, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0007, ANOVA — Week 12 compared to baseline

17. Secondary Outcome: Self-Reported Improvement in the Severity of 'Crepey' Skin on the Neck & Chest
Description: This outcome measures the change in participant-reported scores for the severity of 'crepey' skin on the neck & chest from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of 'crepey' skin severity, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.58 (0.89)
  Week 2 | 2.26 (0.92)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.24 (0.80)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 1.89 (0.91)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 1.81 (0.74)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 1.68 (0.78)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 1.76 (0.76)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.6148, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.7953, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0019, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0008, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0002, ANOVA — Week 12 compared to baseline

18. Secondary Outcome: Self-Reported Improvement in the Severity of Dark Spots on the Skin of the Neck and Chest
Description: This outcome measures the change in participant-reported scores for the severity of dark spots on the skin of the neck and chest from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of dark spot severity, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.89 (0.86)
  Week 2 | 2.21 (1.07)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.14 (0.92)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 1.89 (0.84)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 1.89 (0.88)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 1.84 (0.83)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 1.73 (0.80)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0067, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0055, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

19. Secondary Outcome: Self-Reported Improvement in the Visibility of Fine Lines and Wrinkles on the Skin of the Neck and Chest.
Description: This outcome measures the change in participant-reported scores for the visibility of fine lines and wrinkles on the skin of the neck and chest from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of fine line and wrinkle visibility, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.87 (0.74)
  Week 2 | 2.45 (0.76)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.30 (0.81)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 2.11 (0.88)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 1.97 (0.60)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 2.00 (0.67)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 1.81 (0.81)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.1476, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0106, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0002, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

20. Secondary Outcome: Self-Reported Improvement in the Severity of Sagging on the Neck
Description: This outcome measures the change in participant-reported scores for the severity of sagging on the neck from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of sagging severity, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.55 (0.83)
  Week 2 | 2.18 (0.95)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.00 (0.85)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 1.89 (0.91)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 1.86 (0.79)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 1.81 (0.78)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 1.76 (0.80)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.3224, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0426, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0039, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0040, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0013, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0005, ANOVA — Week 12 compared to baseline

21. Secondary Outcome: Self-Reported Improvement in the Severity of Hyperpigmentation
Description: This outcome measures the change in participant-reported scores for the severity of hyperpigmentation from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of hyperpigmentation, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 3.05 (0.77)
  Week 2 | 2.68 (1.04)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.46 (0.80)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 2.32 (0.82)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 2.16 (0.83)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 2.19 (0.84)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 2.00 (0.82)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.3032, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0237, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0010, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0002, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

22. Secondary Outcome: Self-Reported Improvement in the Visibility of Facial Scars or Blemishes
Description: This outcome measures the change in participant-reported scores for the visibility of facial scars or blemishes from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of scar or blemish visibility, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 2.84 (1.00)
  Week 2 | 2.63 (0.91)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.32 (0.71)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 2.08 (0.76)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 2.14 (0.71)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 1.95 (0.81)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 2.03 (0.83)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p > 0.9999, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.1147, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0016, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0048, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0005, ANOVA — Week 12 compared to baseline

23. Secondary Outcome: Self-Reported Improvement in the Visibility of Any Fine Lines and Wrinkles
Description: This outcome measures the change in participant-reported scores for the visibility of any fine lines and wrinkles from baseline to Week 2, Week 4, Week 6, Week 8, Week 10, and Week 12, using a study-specific questionnaire. Each parameter was scored on a 5-point Likert scale of fine line and wrinkle visibility, including Not noticeable (=1), Barely noticeable (=2), Moderate (=3), Distracting (=4), and Severe (=5). Lower scores indicate greater improvement. This is a negatively weighted item.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | iRESTORE Illumina LED Device Group
Number analyzed (Participants) | 38
Score on a scale
  Baseline | 3.13 (0.66)
  Week 2 | 2.71 (0.87)
  Week 4: number analyzed (Participants) | 37
  Week 4 | 2.51 (0.56)
  Week 6: number analyzed (Participants) | 37
  Week 6 | 2.49 (0.73)
  Week 8: number analyzed (Participants) | 37
  Week 8 | 2.30 (0.70)
  Week 10: number analyzed (Participants) | 37
  Week 10 | 2.24 (0.55)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 2.05 (0.62)
Statistical Analysis 1: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0461, ANOVA — Week 2 compared to baseline
Statistical Analysis 2: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.002, ANOVA — Week 4 compared to baseline
Statistical Analysis 3: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p = 0.0002, ANOVA — Week 6 compared to baseline
Statistical Analysis 4: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 8 compared to baseline
Statistical Analysis 5: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 10 compared to baseline
Statistical Analysis 6: Comparison: iRESTORE Illumina LED Device Group; Test type: Superiority; p < 0.0001, ANOVA — Week 12 compared to baseline

ADVERSE EVENTS:
Time Frame: Participants were asked if they experienced any other effects at the end of the study Week 12.
Arm/Group | iRESTORE Illumina LED Device Group
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 1/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iRESTORE Illumina LED Device Group (N=38)
Dry eyes (Eye disorders) | 1 (1) — One person reported experiencing dry eyes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT07025837/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT07025837/ICF_001.pdf